CLINICAL TRIAL: NCT03285256
Title: Effects of Repeated Memory Training on Memory Function and Addiction Related Processes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants before funding period ended.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00138474
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Substance-Related Disorders
Keywords: Prospective memory, working memory, substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three treatment conditions: an experimental memory training program or one of two comparator memory training programs.
Who Masked: Participant, Investigator
Masking Description: Both the participant and the research assistant conducting the assessments will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Memory Training (Experimental): Experimental memory training program
  Interventions: Behavioral: Experimental memory training
- Comparator Memory Training 1 (Active Comparator): Comparator memory training program
  Interventions: Behavioral: Comparator memory training 1
- Comparator Memory Training 2 (Active Comparator): Alternative comparator memory training program
  Interventions: Behavioral: Comparator memory training 2

INTERVENTIONS:
Behavioral: Experimental memory training — The experimental memory training will be implemented as a computer program that uses state-of-the-art immersive technology to simulate prospective memory in everyday life in which one must remember to carry out tasks throughout the day, while engaging in current ongoing activity. Participants are asked to imagine they have a work-at-home job (ongoing activity), which is an independent program (CogMed QM) designed to train working memory, but that they also need to remember to carry out a number of tasks throughout the day. Using a touch screen, participants will need to touch objects in the simulated environment to appropriately interact with these stimuli according to their pre-assigned tasks.
  Arms: Experimental Memory Training
Behavioral: Comparator memory training 1 — The first comparator memory training intervention will utilize the same overall structure and immersive computer environment as the experimental memory intervention, but will not challenge the same aspects of cognition.
  Arms: Comparator Memory Training 1
Behavioral: Comparator memory training 2 — The second comparator memory training intervention will utilize the same overall structure and immersive computer environment as the experimental memory intervention, but will not challenge the same aspects of cognition.
  Arms: Comparator Memory Training 2

SUMMARY:
Prospective memory is the ability to implement an intention to the future (e.g. remember to take medication, attend a scheduled meeting), and has receive little attention in addiction. The investigators propose that prospective memory plays a critical, yet unrecognized, role in major human behavior change such as that required in addiction treatment. This study will determine the preliminary efficacy of prospective memory training in improving memory and executive functions while reducing illicit drug use in methadone patients. Participants will be randomly assigned to one of three conditions: an experimental memory training program or one of two comparator memory training programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55; provision of written consent
* Enrolled in a substance use treatment program
* Sex with ≥ 2 partners in the last 30 days and sex without a condom on at least one occasion in the last year

Exclusion Criteria:

* Severe psychiatric conditions associated with psychosis or any unstable psychiatric condition
* History of medical, psychiatric, or neurological conditions associated with significant cognitive impairment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in prospective memory over course of training | one month
  Prospective memory will be evaluated within the program itself and measured as the percentage of correct responses within the program. Higher percentages are indicative of greater prospective memory performance.
Change in drug use and substance abuse over course of training. | one month
  Drug use will be evaluated by urinalysis. Negative screens are indicative of drug abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Bayview Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided